CLINICAL TRIAL: NCT04132544
Title: Impact of an Assessment of Risk Factors for Falls and Personalized Care, on Mortality and Institutionalization, After Intervention of the Urgent Medical Assistance Service (SAMU) in the Elderly Person at Home
Brief Title: Risk Factors for Falls After Intervention of the Urgent Medical Assistance Service (SAMU) in the Elderly Person at Home
Acronym: RISING-DOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0453
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2024-05

CONDITIONS: Elderly
Keywords: risks factors; Fall Patients; elderly; Urgent Medical Assistance Service; Emergency Care; 911

STUDY DESIGN:
Intervention Model Description: Interventional multicenter and open, randomized study in parallel groups comparing two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): * a standardized gerontological evaluation (EGS) and a fall balance performed at home or teleconsultation by a Gerontological Assessment Nurse
  * the proposal for a Proposal for a personalized intervention plan (PIP) to correct potentially reversible and modifiable factors
  * a close follow-up by the Gerontological Assessment Nurse for the implementation of the PIP throughout the follow-up period of 24 months (6 home visits and 5 telephone follow-ups).
  Interventions: Other: standardized gerontological evaluation (EGS); Other: Proposal for a personalized intervention plan (PIP); Other: Follow-up
- Comparison group - usual care (Active Comparator): Usual Care with the provision of documentation on simple recommendations for the prevention of falls and aging well.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: standardized gerontological evaluation (EGS) — Evaluation (EGS): initially, the patient benefits from a complete EGS and a complete fall balance realized by a Gerontological Assessment Nurse (initial visit V0) in the 7 working days following the intervention of the SAMU for fall. This assessment is based on the EGS and the assessment of risk factors for falls (HAS, INPES).
  Arms: Intervention group
Other: Proposal for a personalized intervention plan (PIP) — A PIP containing personalized recommendations to improve the patient's state of health, treatment and environment as well as risk factors for falls is proposed during the multi-professional consultation and discussed by telephone with the attending physician (pre-arranged telephone appointment). with the latter).
  The PIP validated by the attending physician is delivered and explained to the patient by the Gerontological Assessment Nurse in the week following the Multidisciplinary Team Meeting (MDTM) during the V1 visit to the patient's home.
  Arms: Intervention group
Other: Follow-up — Four follow-up visits at 6, 12, 18 and 24 months (V2, V3, V4, V5) are performed at the patient's home. During these visits, the Gerontological Assessment Nurse reassesses the person from the gerontological point of view and from the point of view of risk factors for falls.
  A mail containing the elements of interest is sent to the attending physician after each visit. The patient is also contacted by telephone by the Gerontological Assessment Nurse at 2, 4, 9, 15 and 21 months of follow-up to maintain a link, identify possible difficulties and encourage him / her to apply the PIP recommendations.
  Arms: Intervention group
Other: Usual care — The patients included in the "control" group will benefit from the usual care as well as documentation on general recommendations to be put in place to prevent falls and to age in good health [series of brochures published by INPES for the elderly. They are informed by telephone of their home group by the Gerontological Assessment Nurse. The documents are sent by mail to the patient's home address.
  Arms: Comparison group - usual care

SUMMARY:
In this project, the investigators are interested in a particular population, that of elderly subjects who used the SAMU after a fall and who are not hospitalized or are hospitalized less than 24 hours. The scientific literature concerning this population is poor . However, this is a particularly vulnerable population. The Direction of research, studies, evaluation and statistics (DREES) report notes that in 2005 in metropolitan France, 24% of people aged 65 to 75 said they had fallen in the last 12 months. Home falls among seniors may require emergency medical services (EMS).

DETAILED DESCRIPTION:
The first cause of accidental death in people over 65, the fall often has a pejorative impact on the physical, psychological and quality of life . It is also predictive of entry into an institution.

In this project, the investigators propose to evaluate the patient at home with a Gerontological Assessment Nurse working in collaboration with the attending physician, whenever the fall triggers a call to the SAMU (without hospitalization or with hospitalization of less than 24 hours). In addition to the evaluation, the nurse will propose a personalized intervention plan (PIP) based on targeted and prioritized actions.

The Main objective is to study the effect of a personalized intervention plan (PIP) proposed by a Gerontological Assessment Nurse at home in the elderly who used the SAMU for a fall (with on-site care or hospitalization inferior to 24h), on the delay institutionalization or death before institutionalization compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Living at home
* Living at maximum 45 minutes from a hospital center participating in the study (for logistical reasons and practices of study organization)
* Intervention of the SAMU for a fall at home without there being hospitalization or with hospitalization lasting less than 24h
* Patient or trusted person capable of giving telephone information
* Patient or his / her trusted person who has agreed to participate in the study
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Total dependency (ADL at 0)
* Entry in nursing home already scheduled within 3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 952 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The delay between the T0 and Time of occurrence | 2 years
  The composite criterion corresponding to the delay between the T0 and the occurrence of an institutionalization or a death before institutionalization (first event occurring).
  In this pilot study, the average age of subjects was 83.6 years. This is a population for which the goals of home care and delay in the onset of dependence and in the occurrence of death are interesting and feasible.

SECONDARY OUTCOMES:
Number of reminders to the SAMU for fall | 2 years
  The average number of SAMU recalls for drop during the follow-up period will be compared between the two groups at 12 and 24 months after inclusion. This data is collected from a regional database of regulatory data in partnership with the Regional Health Agency (ARS) for all subjects included.
Number of non-programmed hospitalizations | 2 years
  Hospitalizations will be collected for all patients included during the follow-up. We will compare more specifically the unplanned hospitalizations: the average number of unplanned hospitalizations will be compared between the two groups at 12 and 24 months of follow-up.
  This data is collected during the unannounced semi-annual telephone call of the subjects' home groups.
Evolution of the dependence level evaluated by the ADL scale | 2 years
  Katz's scale of functional independence for activities of daily living (Katz S, 1963), commonly known as Katz's ADL (Katz Activity of Living Living Scale), is the most appropriate tool for assessing functional abilities. basic patient. Clinicians generally use this tool to detect problems with performing 6 basic activities of daily living and to plan care accordingly. The score varies from 0 (completely dependent) to 6 (completely autonomous). A score of 4 indicates a moderate functional deficit and 2 a severe functional deficit.
Evolution of the quality-of-life score evaluated by Short Form -12 | 2 years
  The investigators will use the Short Form-12 Quality of Life Scale, which is an abbreviated version of the Medical Outcomes Study Short-Form General Health Survey, with only 12 of the 36 questions that can save a lot of time. It is a generic questionnaire that makes it possible to compare groups of subjects with different pathologies. It measures eight aspects of quality of life that reflect
  World Health Organization (WHO) definition of quality of life: general and mental health, physical and social functioning, physical and emotional health, pain and vitality.
  Compared to the Short Form-36, the Short Form-12 has the advantage of being shorter, less time-consuming, thus easier for the evaluator and better tolerated by patients. Its results are correlated with those of the Short Form-36.
  The Short Form-12 allows to obtain two scores (between 0 and 100, calculated thanks to an algorithm):
  * a score of quality of mental and social life
  * and a physical quality of life score.
Number of deceased or institutionalized subjects | 2 years
  The number of deceased or institutionalized subjects during the follow-up period will be compared between the two groups at 12 and at 24 months of follow-up. This data is collected in both groups during the unannounced semiannual telephone call of the groups belonging to the subjects.
Time to institutionalization | 2 years (up to 54 months for early inclusion)
  The time from T0 to the occurrence of institutionalization will be compared between the two groups until the end of the study (i.e. 54 months for the first patient included). This information will be collected in both groups during the semi-annual follow-up telephone calls, blinded to the participants' group allocation.
Time to death | 2 years (up to 54 months for early inclusion)
  The time from T0 to the occurrence of death will be compared between the two groups until the end of the study (i.e. 54 months for the first patient included). This information will be collected in both groups during the semi-annual follow-up telephone calls, blinded to the participants' group allocation.
  In the event of institutionalization, the clinical research associate will collect the date and cause of death, if applicable, in both groups within the 12 months following admission to a nursing home and/or before the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Fati Nourhashemi, MD, Principal Investigator — University Hospital, Toulouse
Locations (12):
- France (12):
  - CH Albi, Albi
  - CH Cahors, Cahors
  - CH Castres-Mazamet, Castres
  - CHIVA, Foix
  - CH Lannemezan, Lannemezan
  - CH Lavaur, Lavaur
  - CH Montauban, Montauban
  - CH Rodez, Rodez
  - CH Ariège Couserans, Saint-Girons
  - CH Bigorre, Tarbes
  - University Hospital Toulouse, Toulouse
  - Maison de Santé Pluri-professionnelle, Vic-Fezensac

REFERENCES:
- [Result] Bouzid W, Tavassoli N, Berbon C, Qassemi S, Bounes V, Azema O, Shourick J, Nourhashemi F. Impact of a personalised care plan for the elderly calling emergency medical services after a fall at home: The RISING-DOM multi-centre randomised controlled trial protocol. BMC Geriatr. 2022 Mar 4;22(1):182. doi: 10.1186/s12877-022-02850-w. PMID 35246053
- [Result] Bouzid W, Tavassoli N, Berbon C, Qassemi S, Vaysset S, Poly M, Bounes V, Shourick J, Nourhashemi F. Exploring Population Characteristics and Recruitment Challenges in Older People Experiencing Falls at Home without Hospitalization or with an Emergency Department Visit: Insights from the RISING-DOM Experience. Clin Interv Aging. 2023 Dec 1;18:1995-2008. doi: 10.2147/CIA.S421053. eCollection 2023. PMID 38058551
- [Result] Ailliaud A, Moulis E, Vaysset S, Berbon C, Tavassoli N, Bouzid W, Oliveira Soares C, Qassemi S, Nourashemi F. [Assessment in the home of the elderly following a first fall with Samu intervention]. Soins Gerontol. 2022 Jan-Feb;27(153):23-25. doi: 10.1016/j.sger.2021.11.008. Epub 2021 Nov 24. French. PMID 35120719